CLINICAL TRIAL: NCT04943263
Title: A Comparison of Body Temperature Measured From the Cuff Surface of the Endotracheal Tube and Core Temperature in Living Donor Liver Transplantation
Brief Title: A Comparison of Temperature Measurement During Living Donor Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Oneclickmedical Co., Ltd. (Seoul, South Korea) (Unknown)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20210623
Record Dates: First submitted 2021-06-23; First posted 2021-06-29 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Living Donor Liver Transplantation
Keywords: core temperature; esophageal temperature; tracheal temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracheal Temperature (Experimental): Intubation done with a temperature sensor located on the cuff surface of the endotracheal tube
  Interventions: Other: Tracheal Temperature

INTERVENTIONS:
Other: Tracheal Temperature — Temperature measured from the endotracheal tube compared with the esophageal temperature

SUMMARY:
The purpose of this study is to compare the temperature measured from the cuff surface of the endotracheal tube and core temperature measured at the esophagus in living donor liver transplantation recipients.

DETAILED DESCRIPTION:
Hypothermia occurs frequently in patients undergoing surgery and is known to be related with many postoperative complications. Patients undergoing living donor liver transplantation are usually monitored using an esophageal stethoscope. However, because patients with liver cirrhosis have the risk of variceal bleeding, placement of an esophageal stethoscope can increase the risk of bleeding.

There have been previous reports that temperature monitoring at the cuff surface of an endotracheal tube is not only safe but also provides accurate and reliable data during mild hypothermia after cardiac arrest.

This study compares the temperature measured from the cuff surface of the endotracheal tube and core temperature measured at the esophagus and additionally core temperature measured by a pulmonary artery catheter. The study participants are intubated with an endotracheal tube that has a temperature sensor at the cuff surface of the tube. The rest of the procedure is done according to Seoul National University Hospital's protocol for liver transplantation: an esophageal stethoscope is placed for temperature monitoring and a central line is placed with a Multi-Access lumen Catheter and a pulmonary artery catheter is placed. The temperature measurements from the endotracheal tube and measurements from the esophageal stethoscope are compared at the following 5 phases: 1. preanhepatic phase, 2. anhepatic phase 1 (recipient hepatectomy - IVC clamping), 3. anhepatic phase 2 (IVC clamping - reperfusion), 4. Reperfusion phase, 5. Neohepatic phase.

ELIGIBILITY:
Inclusion Criteria:

* routine living donor liver transplantation recipients needing pulmonary artery catheterization who have been informed and given consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-08-13 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of temperature from the cuff surface of the endotracheal tube and esophageal temperature | Phase 1 (preanhepatic): 60 minutes after the anesthetic induction
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and esophageal temperature | Phase 2 (anhepatic 1): 10 minutes after recipient hepatectomy
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and esophageal temperature | Phase 3 (anhepatic 2): 10 minutes after IVC clamping
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and esophageal temperature | Phase 4 (Reperfusion): 5 minutes after Reperfusion
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and esophageal temperature | Phase 5 (neohepatic): 1 hour after Reperfusion
  temperature

SECONDARY OUTCOMES:
Comparison of temperature from the cuff surface of the endotracheal tube and temperature measured at the pulmonary artery catheter | Phase 1 (preanhepatic): 60 minutes after the anesthetic induction
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and temperature measured at the pulmonary artery catheter | Phase 2 (anhepatic 1): 10 minutes after recipient hepatectomy
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and temperature measured at the pulmonary artery catheter | Phase 3 (anhepatic 2): 10 minutes after IVC clamping
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and temperature measured at the pulmonary artery catheter | Phase 4 (Reperfusion): 5 minutes after Reperfusion
  temperature
Comparison of temperature from the cuff surface of the endotracheal tube and temperature measured at the pulmonary artery catheter | Phase 5 (neohepatic): 1 hour after Reperfusion
  temperature

CONTACTS AND LOCATIONS:
Overall Officials: Hee Soo Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Lefrant JY, Muller L, de La Coussaye JE, Benbabaali M, Lebris C, Zeitoun N, Mari C, Saissi G, Ripart J, Eledjam JJ. Temperature measurement in intensive care patients: comparison of urinary bladder, oesophageal, rectal, axillary, and inguinal methods versus pulmonary artery core method. Intensive Care Med. 2003 Mar;29(3):414-8. doi: 10.1007/s00134-002-1619-5. Epub 2003 Feb 8. PMID 12577157
- [Background] Erickson RS, Kirklin SK. Comparison of ear-based, bladder, oral, and axillary methods for core temperature measurement. Crit Care Med. 1993 Oct;21(10):1528-34. doi: 10.1097/00003246-199310000-00022. PMID 8403963
- [Background] Yamakage M, Kawana S, Watanabe H, Namiki A. The utility of tracheal temperature monitoring. Anesth Analg. 1993 Apr;76(4):795-9. doi: 10.1213/00000539-199304000-00020. PMID 8466020
- [Background] Torossian A. Thermal management during anaesthesia and thermoregulation standards for the prevention of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):659-68. doi: 10.1016/j.bpa.2008.07.006. PMID 19137809
- [Background] Hayes JK, Collette DJ, Peters JL, Smith KW. Monitoring body-core temperature from the trachea: comparison between pulmonary artery, tympanic, esophageal, and rectal temperatures. J Clin Monit. 1996 May;12(3):261-9. doi: 10.1007/BF00857648. PMID 8823651
- [Background] Haugk M, Stratil P, Sterz F, Krizanac D, Testori C, Uray T, Koller J, Behringer W, Holzer M, Herkner H. Temperature monitored on the cuff surface of an endotracheal tube reflects body temperature. Crit Care Med. 2010 Jul;38(7):1569-73. doi: 10.1097/CCM.0b013e3181e47a20. PMID 20495450
- [Background] Sun Y, Jia LL, Yu WL, Yu HL, Sheng MW, Du HY. The changes of intraoperative body temperature in adult liver transplantation: A retrospective study. Hepatobiliary Pancreat Dis Int. 2018 Dec;17(6):496-501. doi: 10.1016/j.hbpd.2018.08.006. Epub 2018 Aug 29. PMID 30205926